CLINICAL TRIAL: NCT07125339
Title: High-resolution Magnetic Resonance Vessel Wall Imaging of Intracranial and Extracranial Plaques: a Prospective Cohort Registration Study
Brief Title: High-resolution Magnetic Resonance Vessel Wall Imaging of Plaques
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: HELP Study
Record Dates: First submitted 2025-08-06; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Atherosclerotic Stenosis
Keywords: high resolution vessel wall imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke group: Patients with moderate to severe stenosis (stenosis degree: 50% ~ 99%) in both intracranial and extracranial arteries were considered for enrollment in this study.

SUMMARY:
The primary objective of this study is to investigate the predictive value of High-resolution magnetic resonance vessel wall imaging for future stroke occurrence in patients with moderate to severe intracranial and extracranial artery stenosis.

The secondary objective is to explore the predictive value of baseline high-resolution magnetic resonance vessel wall imaging for plaque progression.

DETAILED DESCRIPTION:
Carotid artery origin and intracranial atherosclerotic stenosis (ICAS) are among the leading causes of ischemic cerebrovascular events worldwide, with ICAS accounting for up to 46.6% of ischemic stroke or transient ischemic attacks (TIA) cases in China. Vascular imaging-defined lumen narrowing and clinical manifestations have long been recognized as primary contributors to subsequent ischemic cerebrovascular events. While it is widely accepted that most ischemic events result from ruptured atherosclerotic plaques, hemodynamic disturbances caused by plaque progression within and beyond the cranium, collateral or perforator occlusions, and distal embolism from plaque detachment also play significant roles. Current clinical decision-making relying solely on lumen narrowing dimensions presents substantial limitations. Compared to lumen narrowing alone, detailed characterization of plaque morphology and composition correlates more closely with clinical presentations and subsequent ischemic events.

Advanced high-resolution vessel wall imaging (HR-VWI) technology has achieved 2D and 3D imaging of intracranial and extracranial arterial walls. By suppressing blood flow within the vessels, it can clearly display the morphology and signal characteristics of the vascular walls: Non-invasively describe the detailed structure of atherosclerosis, identifying plaque components, enhancement intensity, reconstruction type, and load, while evaluating the characteristics of vulnerable plaques in extracranial carotid arteries and ICAS, such as intraplaque hemorrhage (IPH), lipid-rich necrotic core (LRNC), and ulcers. Previous studies have shown that these plaque features can provide additional value for distinguishing between stroke cases and asymptomatic patients with narrowed arteries.

However, most of these studies are cross-sectional in nature, and due to limited data, their conclusions vary. Some reports suggest that symptomatic ICAS patients with plaque enhancement may be more related to future ischemic events, while other studies argue that the correlation is minimal. Additionally, previous research investigating the temporal changes in plaque characteristics and their relationship with recurrent stroke has been constrained by small sample sizes (N <15), leading to inconclusive conclusions.

Therefore, more comprehensive studies are needed to evaluate the value of baseline HR-VWI in identifying patients with intracranial and extracranial arterial stenosis at risk of ischemic cerebrovascular events in the future. Through wall plaque imaging studies, it is expected that multi-modal imaging can be used to stratify stroke risk based on cerebral vascular plaques.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Medium or severe stenosis of the internal carotid artery, middle cerebral artery, V4 segment of vertebral artery or basilar artery [stenosis degree: 50% ~ 99%, confirmed by CTA, MRA or DSA];
* Accept high resolution magnetic resonance angiography; The patient or the legal representative of the patient is able and willing to sign an informed consent form

Exclusion Criteria:

* Non-atherosclerotic intracranial and extracranial artery stenosis, such as dissection, smoke disease, etc.;
* There are contraindications to MRI, such as claustrophobia, metal implants, etc.;
* Renal insufficiency, elevated serum creatinine (more than twice the upper limit of normal);
* Patients with severe cardiopulmonary diseases were considered unsuitable for this study;
* Gadolinium contrast agent allergy;
* Participants who were unable to complete the study due to mental illness, cognitive or emotional disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe stenosis (stenosis degree: 50% ~ 99%) in both intracranial and extracranial arteries were considered for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 605 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Lumen Stenosis Rate | 2024.08-2027.12
  The lumen stenosis rate is calculated using the 3D TOF-MRA measurement of the vertebral-basilar artery's narrowest diameter and the normal diameter at the proximal end. The calculation follows the Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) standard formula: Lumen Stenosis Rate = [1- (Narrowest Diameter / Normal Diameter at Proximal End)] × 100%
Identify different plaque components | 2024.08-2027.12

SECONDARY OUTCOMES:
Ejection index and maximum wall thickness | 2024.08-2027.12
  Select the narrowest lumen level and manually outline the lumen and wall boundary at the narrowest point. Ejection index = (maximum wall thickness-minimum wall thickness)/ maximum wall thickness
Wall thickness | 2024.08-2027.12
  maximum wall thickness, minimum wall thickness and average wall thickness
Patch load | 2024.08-2027.12
  Select the narrowest lumen level and manually outline the lumen and wall boundaries at the narrowest point. Mainly measure the lumen area (LA), wall area (WA), and normalized wall index (NWI). NWI = WA / (WA + LA) × 100%
Vascular reconstruction index RR | 2024.08-2027.12
  measured by the ratio of the outer wall area of the blood vessel in the lesion to that of the adjacent normal blood vessel
Plaque-to-pituitary stalk contrast enhancement ratio (CR) | 2024.08-2027.12
  CR = (SI plaque post / SI stalk post) × 100%; signal intensity (signal intensity, SI)

CONTACTS AND LOCATIONS:
Overall Officials: Yueqi Zhu, MD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No